CLINICAL TRIAL: NCT05695885
Title: Stepped Transition in Education Program for Emerging Adults With Autism: Pilot Effectiveness Trial
Brief Title: STEPS Implementation Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama, Tuscaloosa (Other)
Responsible Party: Principal Investigator, Susan White, Professor, University of Alabama, Tuscaloosa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 22-07-5746
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Autism Spectrum Disorder
Keywords: transition; adulthood; employment; education
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Parallel RCT
Who Masked: Outcomes Assessor
Masking Description: The main outcome measure is completed by a trained evaluator unaware of assigned treatment condition (i.e., the Independent Evaluator; IE).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STEPS (Experimental): 14 session counseling targeting adult independence skills
  Interventions: Behavioral: STEPS
- Control (Other): Services as usual
  Interventions: Behavioral: Services as usual (SAU)

INTERVENTIONS:
Behavioral: STEPS — behavioral counseling
  Arms: STEPS
Behavioral: Services as usual (SAU) — behavioral counseling normally provided
  Arms: Control

SUMMARY:
This study will inform understanding of how to support emerging adults with autism spectrum disorder (ASD). The investigators will use a theoretically informed and research-based transition support program developed for people with ASD and test how effective it is when delivered by community agencies. Results will provide information on the effectiveness of the program as well as on mechanisms of change and contextual factors that promote or impede implementation.

DETAILED DESCRIPTION:
The long-term goal of this research is to improve adult outcomes for people with autism spectrum disorder (ASD). Autistic adolescents and young adults tend to have worse outcomes with respect to employment, education, and quality of life, than neurotypical peers. These outcomes include under-enrollment into college, unemployment, and limited functional independence. Research-informed transition planning that addresses core impairments in skills related to adult autonomy, including self-knowledge, self-determination, and self-regulation, may improve outcomes for this growing population. In prior research, investigators developed a stakeholder involved transition program (STEPS) and found it to be feasible, acceptable, and efficacious. Data from a small randomized controlled trial (RCT) focusing on feasibility indicated that it was acceptable to participants and suggested STEPS was effective in improving readiness for transition to adulthood. The team will now test the effectiveness of STEPS, and engagement of target mechanisms, in partnership with four community agencies. This study is designed as a Hybrid Type 1, which focuses primarily on intervention effectiveness with a secondary focus on factors related to implementation. Immediate (post-treatment) and longer-term (six month follow-up) clinical outcomes of adult functional outcomes and vocational engagement will be assessed. The degree to which STEPS leads to change in the theoretical mediating mechanisms (i.e., adult autonomy skills) will be examined, as well as a formal test of mediation (i.e., the degree to which change in adult autonomy skills leads to change in adult functional outcomes). Providers will provide qualitative information on implementation such as thoughts on STEPS' cultural sensitivity, and quantitative data on the appropriateness, feasibility, and acceptability of STEPS. Providers' sustained use of STEPS with clients in the six months after study enrollment has ended will also be tracked. This research will produce findings that have the potential to shift clinical practice related to transition to adulthood for people with ASD. In light of the fact that approximately 70,000 people with ASD age into adulthood every year and the economic burden associated with ASD, the potential public health impact of this research is considerable.

ELIGIBILITY:
Inclusion Criteria:

* 16-25 years of age
* have confirmed diagnosis of ASD
* want to participate in STEPS
* have a caregiver/parent who can complete assessments

Exclusion Criteria:

* presence of suicidal/homicidal intent

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Transition Readiness Scale-Revised | 30 days
  This caregiver and self-report questionnaire has a range of possible scores from 30 to 120, with higher scores indicating greater readiness.assigned condition. Scores are categorical in nature: 0 = no evidence of progression toward goals, 1 = some evidence, 2 = strong evidence of progression toward goals.

SECONDARY OUTCOMES:
Relationships, Employment, Autonomy, and Life Satisfaction | 30 days
  This is a questionnaire completed by caregiver and participant. Higher scores indicate greater autonomy, independence, and satisfaction. On the self-report measure scores range as follows for Frequency: social engagement (0-56), outside meaningful activities (0-32), self-care (0-88), independence (0-56), and romance (0-16) and level of support ranges are: social engagement (0-68), outside meaningful activities (0-32), self-care (0-76), independence (0-48), finances (0-12), and satisfaction (0-132). On caregiver-report, frequency subscales range as follows: degree of social contact (0-28), social initiation (0-60), work/finances (0-64), autonomy (0-56), care of self and home (0-72), and support subscales range as follows: social engagement (0-68), self-care (0-144), work activity (0-28), independence (0-16), and finances (0-24).
Rehabilitation Success | 30 days
  This brief interview on progress made toward educational or employment goals is completed with participant and caregiver, conducted by an examiner unaware of assigned condition. Scores are categorical in nature: 0 = no evidence of progress toward goals, 1 = some evidence of progress toward goals, 2 = moderate evidence of progress toward goals, and 3 = clear strong evidence of progress toward goals. Higher scores indicate greater goal attainment.

CONTACTS AND LOCATIONS:
Locations (1):
- Center o=for Youth Development and Intervention, Tuscaloosa, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
we submit de-identified data to NIH repository (NDA)
Supporting Information: Study Protocol
Time Frame: one year after study closure